CLINICAL TRIAL: NCT05197595
Title: Efficacy of a Compassion Program for the Reduction of Psychological Distress in University Students
Brief Title: Efficacy of a Compassion Program in University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18/2021
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Wellness
Keywords: Attachment-based compassion therapy; Students; Psychological well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassion condition (Experimental): 90-minute group sessions, held once a week over a space of 6 weeks, and is offered as an extra-curricular activity.
  Interventions: Behavioral: Attachment-based compassion therapy
- Relaxation condition (Active Comparator): 90-minute group sessions, held once a week over a space of 6 weeks, and will be offered as an extracurricular activity.
  Interventions: Behavioral: Relaxation program

INTERVENTIONS:
Behavioral: Attachment-based compassion therapy — Compassion program consists of 6 sessions of 90 minutes/session (15-20 people) Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months
  Arms: Compassion condition
Behavioral: Relaxation program — Relaxation program consists of 6 sessions of 90 minutes/session (15-20 people) Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months
  Arms: Relaxation condition

SUMMARY:
University life is a challenging period. College students are exposed to a large number of stressors such as increased workload, multitasking, new responsibilities, changes in sleep and eating habits, social stressors, financial concerns and future employability, unlimited access to technology, etc. The participation of some of them in unhealthy activities should also be noted.

There is sufficient evidence to affirm that high levels of stress cause different alterations in students, such as attention and concentration deficits, difficulties in memorizing and solving problems, low productivity and poor academic performance. Due to this, in addition to the psychological and social impact of said mental health problems, the academic functioning of the students decreases and the dropout rates increase, which represents a problem for themselves and for the institutions. On the other hand, students and future professionals in training run the risk of suffering burnout as a consequence of the chronic stress to which they are subjected, with the consequent negative effects on their future professional practice.

The main objective of the present research is to evaluate the efficacy of a six-week compassion program for the reduction of psychological distress in university students compared to an active control condition based on relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30 years old.
* Study undergraduate or master's degrees at the University of Zaragoza.
* Understand perfectly spoken and written Spanish.
* Grant informed consent.

Exclusion Criteria:

* Any diagnose of disease that may affect central nervous system (brain pathology traumatic brain injury, dementia, etc.).
* Other psychiatric diagnoses or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders, etc.) except for anxious pathology or personality disorders.
* Any medical, infectious or degenerative disease that may affect mood, presence of delusional ideas or hallucinations consistent or not with mood, and suicide risk.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-06 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale - 21 (DASS-21) | Baseline
  In the compassion program group
Depression Anxiety and Stress Scale - 21 (DASS-21) | Baseline
  In the relaxation program group
Depression Anxiety and Stress Scale - 21 (DASS-21) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Depression Anxiety and Stress Scale - 21 (DASS-21) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Depression Anxiety and Stress Scale - 21 (DASS-21) | Six-months follow-up
  In the compassion condition group
Depression Anxiety and Stress Scale - 21 (DASS-21) | Six-months follow-up
  In the relaxation program group

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the compassion condition group
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the relaxation program group
Positive and negative affect (PANAS) | Baseline
  In the compassion condition group
Positive and negative affect (PANAS) | Baseline
  In the relaxation program group
Positive and negative affect (PANAS) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Positive and negative affect (PANAS) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Positive and negative affect (PANAS) | Six-months follow-up
  In the compassion condition group
Positive and negative affect (PANAS) | Six-months follow-up
  In the relaxation program group
Emotional Regulation Questionnaire (ERQ) | Baseline
  In the compassion condition group
Emotional Regulation Questionnaire (ERQ) | Baseline
  In the relaxation program group
Emotional Regulation Questionnaire (ERQ) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Emotional Regulation Questionnaire (ERQ) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Emotional Regulation Questionnaire (ERQ) | Six-months follow-up
  In the compassion condition group
Emotional Regulation Questionnaire (ERQ) | Six-months follow-up
  In the relaxation program group
Maslach Burnout Inventory Student Survey (MBI-SS) | Baseline
  In the compassion condition group
Maslach Burnout Inventory Student Survey (MBI-SS) | Baseline
  In the relaxation program group
Maslach Burnout Inventory Student Survey (MBI-SS) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Maslach Burnout Inventory Student Survey (MBI-SS) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Maslach Burnout Inventory Student Survey (MBI-SS) | Six-months follow-up
  In the compassion condition group
Maslach Burnout Inventory Student Survey (MBI-SS) | Six-months follow-up
  In the relaxation program group

OTHER OUTCOMES:
The Relationship Questionnaire (RQ) | Baseline
  In the compassion condition group
The Relationship Questionnaire (RQ) | Baseline
  In the relaxation program group
The Relationship Questionnaire (RQ) | Post-treatment 6 weeks from baseline
  In the compassion condition group
The Relationship Questionnaire (RQ) | Post-treatment 6 weeks from baseline
  In the relaxation program group
The Relationship Questionnaire (RQ) | Six-months follow-up
  In the compassion condition group
The Relationship Questionnaire (RQ) | Six-months follow-up
  In the relaxation program group
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline
  In the compassion condition group
Acceptance and Action Questionnaire-II (AAQ-II) | Baseline
  In the relaxation program group
Acceptance and Action Questionnaire-II (AAQ-II) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Acceptance and Action Questionnaire-II (AAQ-II) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Acceptance and Action Questionnaire-II (AAQ-II) | Six-months follow-up
  In the compassion condition group
Acceptance and Action Questionnaire-II (AAQ-II) | Six-months follow-up
  In the relaxation program group
Sussex-Oxford Compassion for Others Scale & SussexOxford Compassion for the Self Scale (SOCS) | Baseline
  In the compassion condition group
Sussex-Oxford Compassion for Others Scale & SussexOxford Compassion for the Self Scale (SOCS) | Baseline
  In the relaxation program group
Sussex-Oxford Compassion for Others Scale & SussexOxford Compassion for the Self Scale (SOCS) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Sussex-Oxford Compassion for Others Scale & SussexOxford Compassion for the Self Scale (SOCS) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Sussex-Oxford Compassion for Others Scale & SussexOxford Compassion for the Self Scale (SOCS) | Six-months follow-up
  In the compassion condition group
Sussex-Oxford Compassion for Others Scale & SussexOxford Compassion for the Self Scale (SOCS) | Six-months follow-up
  In the relaxation program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Baseline
  In the compassion condition group
Five Facets of Mindfulness Questionnaire (FFMQ) | Baseline
  In the relaxation program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Post-treatment 6 weeks from baseline
  In the compassion condition group
Five Facets of Mindfulness Questionnaire (FFMQ) | Post-treatment 6 weeks from baseline
  In the relaxation program group
Five Facets of Mindfulness Questionnaire (FFMQ) | Six-months follow-up
  In the compassion condition group
Five Facets of Mindfulness Questionnaire (FFMQ) | Six-months follow-up
  In the relaxation program group

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Servet University Hospital, Zaragoza, Spain

REFERENCES:
- [Derived] Beltran-Ruiz M, Fernandez S, Garcia-Campayo J, Puebla-Guedea M, Lopez-Del-Hoyo Y, Navarro-Gil M, Montero-Marin J. Effectiveness of attachment-based compassion therapy to reduce psychological distress in university students: a randomised controlled trial protocol. Front Psychol. 2023 Aug 24;14:1185445. doi: 10.3389/fpsyg.2023.1185445. eCollection 2023. PMID 37691796